CLINICAL TRIAL: NCT01545908
Title: A Randomized Controlled Trial of Fecal Biotherapy for the Induction of Remission in Active Ulcerative Colitis
Brief Title: Fecal Biotherapy for the Induction of Remission in Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Paul Moayyedi, Director, Division of Gastroenterology, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REB # 11-600
Record Dates: First submitted 2012-02-22; First posted 2012-03-07 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Ulcerative Colitis
Keywords: Fecal transplant; induction of remission; active ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo enema (Placebo Comparator): Participants in this arm undergo 6 retention enemas, week 1, week 2, week 3, week 4, week 5, week 6
  Interventions: Other: Placebo enema
- Fecal transplant from an unrelated donor (Active Comparator): Participants in this arm undergo 6 retention enemas,week 1, week 2, week 3, week 4, week 5, week 6,using stool specimen prepared from a healthy, screened donor.
  Interventions: Other: Fecal transplant

INTERVENTIONS:
Other: Fecal transplant — Participants in this arm undergo 6 retention enemas,using stool specimen prepared from a healthy, screened unrelated donor.
  Other Names: Fecal bacteriotherapy, fecal biotherapy.
  Arms: Fecal transplant from an unrelated donor
Other: Placebo enema — Patients will receive placebo enema, week 1, week 2, week 3, week 4, week 5, week 6
  Other Names: saline enema
  Arms: placebo enema

SUMMARY:
Ulcerative colitis is a condition that mainly affects young adults where the lining of the bowel is inflamed causing bloody diarrhea. The cause of ulcerative colitis is unknown and treatments remain imperfect with no cure for the disease. Initial success has been shown with a highly novel treatment where patients with active ulcerative colitis receive a fecal enema to try and replace their stool containing bacteria that may be driving their disease with that from a healthy donor. To assess if this works by comparing how well it treats the disease compared to a placebo enema.

DETAILED DESCRIPTION:
Hypothesis Fecal biotherapy will be more effective than placebo at inducing remission in patients with active UC.

Approach and work plan Patients aged 18 or over with active UC defined as a Mayo score (13) more than 3 with an endoscopic score more than 0 will be eligible for the study. Subjects will be excluded if they are participating in another clinical trial, are unable to give informed consent, have severe comorbid medical illness, have concomitant Clostridium difficile infection or have severe UC requiring hospitalization. Continued treatment with 5-ASA, azathioprine, 6-mercaptopurine or anti-TNF therapy (e.g. infliximab) will be permitted if taken at stable dose for more or equal to 12 weeks prior to randomization. Eligible patients will be randomized to receive fecal biotherapy or placebo. Fecal biotherapy will be provided by an unrelated donor who is able to give informed consent, travel to the treatment centre at St Joseph's Hospital, Hamilton and able to collect fecal sample as needed for the fecal transplantation protocol. Fecal microbiome profiling will be carried out using both Roche 454 pyrosequencing and Illumina sequencing.

One hundred and thirty active UC patients will be randomized 1:1 according to a computer generated randomization list. Randomization will be administered centrally at the GI Clinical Trials Unit to ensure concealment of allocation. Eligible patients will be randomized to receive a weekly fecal biotherapy enema or a placebo enema for six weeks. In order to mitigate a placebo effect, both the patient and study staff will be blinded to the allocation of the treatment. An unblinded, independent laboratory technologist will prepare the retention enema according to the treatment arm to which the patient is assigned. The enema containers will be fully colour-tinted from the tip to the bottom of the container. The container will be placed inside a paper bag, which contains baking soda to absorb the odor. Both the patient and the study nurse will be required to wear a tightly fitted mask at all times during the infusion and retention of the enema.

Subjects will have a sigmoidoscopy (or colonoscopy if clinically indicated), physician assessment and complete a Mayo score (13) and IBDQ questionnaire (15) at baseline. The physician assessment, IBDQ and partial Mayo score (Mayo score without the sigmoidoscopy) will be repeated at 3 weeks. A repeat sigmoidoscopy, physician assessment IBDQ and Mayo score will be completed at 6 weeks, at exit from the study. No new medical therapies (e.g. corticosteroids, antibiotics, probiotics) will be permitted during the six-week study period. At the end of the treatment component of the study, fecal biotherapy will be offered to the participants in the placebo arm with clinical and sigmoidoscopic evidence of active UC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or over with active UC defined as a Mayo score (13) more than 3 with an endoscopic score more than 0 will be eligible for the study
* Continued treatment with 5-ASA, azathioprine, 6-mercaptopurine or anti-TNF therapy (e.g. infliximab) will be permitted if taken at stable dose for more than or equal to 12 weeks prior to randomization.

Exclusion Criteria:

* Subjects will be excluded if they are participating in another clinical trial, are unable to give informed consent, have severe comorbid medical illness, have concomitant Clostridium difficile infection or have severe UC requiring hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the randomized trial will remission of UC with colonic mucosa healing defined as Mayo endoscopy score = 0 at 6 weeks | Subjects will have a sigmoidoscopy, physician assessment and complete a Mayo score and IBDQ questionnaire at baseline, week 3 (no sigmoidoscopy is required), week 6 at exit from the study.
  All analyses will be conducted using both intention-to-treat and per-protocol, and the differences in remission rates and relapse rates between the two groups will be statistically analysed. The usual descriptive statistics using Fisher exact test, proportion test, rank test and t-test will be used to compare the two populations making sure that the randomization split the sample into two homogenous sub-samples. Logistic regression and estimating equations will also be used.

SECONDARY OUTCOMES:
Secondary outcomes include endoscopic and clinical remission defined as a Mayo score = 0 and improvement in symptoms defined as a decrease ≥3 in the Mayo score from baseline at 6 weeks. | Subjects will have a sigmoidoscopy, physician assessment and complete a Mayo score and IBDQ questionnaire at baseline, week 3 (no sigmoidoscopy is required), week 6 at exit from the study.
  All analyses will be conducted using both intention-to-treat and per-protocol, and the differences in remission rates and relapse rates between the two groups will be statistically analysed. The usual descriptive statistics using Fisher exact test, proportion test, rank test and t-test will be used to compare the two populations making sure that the randomization split the sample into two homogenous sub-samples. Logistic regression and estimating equations will also be used.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lee, MD, Principal Investigator — St. Joseph's Hamilton Healthcare; Paul Moayyedi, MD, FRCP, Principal Investigator — Hamilton Health Sciences, McMaster University
Locations (2):
- Canada (2):
  - Hamilton Health Sciences / McMaster University, Hamilton, Ontario
  - St. Joseph's Hamilton Healthcare, Hamilton, Ontario

REFERENCES:
- [Result] Bakken JS, Borody T, Brandt LJ, Brill JV, Demarco DC, Franzos MA, Kelly C, Khoruts A, Louie T, Martinelli LP, Moore TA, Russell G, Surawicz C; Fecal Microbiota Transplantation Workgroup. Treating Clostridium difficile infection with fecal microbiota transplantation. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1044-9. doi: 10.1016/j.cgh.2011.08.014. Epub 2011 Aug 24. PMID 21871249
- [Derived] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665